CLINICAL TRIAL: NCT05263921
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF PF-07321332/RITONAVIR ORAL POWDER IN 3 DIFFERENT DELIVERY VEHICLES RELATIVE TO THE COMMERCIAL PF-07321332/RITONAVIR TABLETS IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITIONS
Brief Title: Relative Bioavailability Study of PF-07321332/Ritonavir Oral Powder Relative to the Commercial Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671024
Record Dates: First submitted 2022-02-25; First posted 2022-03-03 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Bioavailability
Keywords: coronavirus disease 2019 (COVID-19); severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nirmatrelvir
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: PF-07321332/ritonavir (Active Comparator): PF-07321332 ritonavir
  Interventions: Drug: PF-07321332/ritonavir
- Treatment B: PF-07321332/ritonavir (Experimental): PF-07321332/ritonavir mixed with water
  Interventions: Drug: PF-07321332/ritonavir
- Treatment C: PF-07321332/ritonavir (Experimental): PF-07321332/ritonavir mixed with applesauce
  Interventions: Drug: PF-07321332/ritonavir
- Treatment D: PF-07321332/ritonavir (Experimental): PF-07321332/ritonavir mixed with vanilla pudding
  Interventions: Drug: PF-07321332/ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — Single oral dose of PF-07321332/ritonavir under fasted conditions
  Arms: Treatment A: PF-07321332/ritonavir
Drug: PF-07321332/ritonavir — Single oral dose of PF-07321332/ritonavir mixed with water under fasted conditions
  Arms: Treatment B: PF-07321332/ritonavir
Drug: PF-07321332/ritonavir — Single oral dose of PF-07321332/ritonavir mixed with applesauce under fasted conditions
  Arms: Treatment C: PF-07321332/ritonavir
Drug: PF-07321332/ritonavir — Single oral dose of PF-07321332/ritonavir mixed with vanilla pudding under fasted conditions
  Arms: Treatment D: PF-07321332/ritonavir

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of PF-07321332/ritonavir oral powder relative to the commercial tablet formulation under fasted condition in healthy adult participants. The study will also assess the effect of 3 different food vehicles on the relative bioavailability of the PF-07321332/ritonavir oral powder formulation as well as the safety, tolerability, and palatability of PF-07321332/ritonavir oral powder in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination (PE), laboratory tests, vital signs and standard 12 lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a phase 1, open label, single dose, randomized, crossover study in healthy adult participants. A total of 12 participants were assigned to the study, participating in 4 study periods to receive 4 different treatments, and 11 participants completed the study and 1 participant discontinued from the study intervention due to family emergency.
Groups:
- Sequence 1: Treatment A-> B-> C-> D; Sequence 2: Treatment B-> D-> A-> C; Sequence 3: Treatment C-> A-> D-> B; Sequence 4: Treatment D-> C-> B-> A: Treatment A: Nirmatrelvir/ritonavir 300/100 mg commercial tablets. Treatment B: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with water. Treatment C: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with applesauce.
  Treatment D: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding.
  All treatments were administered under fasted conditions, and a minimum of 4-day washout was planned between each treatment.
Period: Overall Study
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> D-> A-> C | Sequence 3: Treatment C-> A-> D-> B | Sequence 4: Treatment D-> C-> B-> A
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Other: family emergency. | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Participant
Groups:
- All Participants: All participants enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Number analyzed (Participant) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.25 (12.800)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCinf of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: Area under the plasma concentration time profile from time 0 extrapolated to infinity (AUCinf) was measured. AUCinf was determined by AUClast + (Clast/kel), where Clast is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets: Nirmatrelvir/ritonavir 300/100 mg commercial tablets were administered under fasted conditions.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with water were administered under fasted conditions.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with applesauce were administered under fasted conditions.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding were administered under fasted conditions.
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
nanogram*hour per milliliter (ng*hr/mL) | 28670 (36) | 30780 (25) | 33170 (33) | 36020 (27)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; Reference: Nirmatrelvir/ritonavir 300/100 mg commercial tablets; Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with water; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 107.35, 90% CI 2-sided [99.66 to 115.64]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; Reference: Nirmatrelvir/ritonavir 300/100 mg commercial tablets Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with applesauce; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 120.73, 90% CI 2-sided [112.09 to 130.03]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; Reference: Nirmatrelvir/ritonavir 300/100 mg commercial tablets Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 125.04, 90% CI 2-sided [116.08 to 134.69]

2. Primary Outcome: AUClast of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: Area under the plasma concentration time profile from time 0 to the time of the last quantifiable concentration (Clast) was measured. AUClast was determined by Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
ng*hr/mL | 27790 (36) | 30230 (27) | 32180 (33) | 35580 (27)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; [analysis description as in outcome 1, analysis 1]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 108.80, 90% CI 2-sided [101.06 to 117.14]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; [analysis description as in outcome 1, analysis 2]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 120.95, 90% CI 2-sided [112.36 to 130.20]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; [analysis description as in outcome 1, analysis 3]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 127.39, 90% CI 2-sided [118.32 to 137.15]

3. Primary Outcome: Cmax of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: Maximum plasma concentration (Cmax) was measured. Cmax was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
nanogram per milliliter (ng/mL) | 2817 (31) | 3254 (23) | 4025 (22) | 4572 (19)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; [analysis description as in outcome 1, analysis 1]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 115.10, 90% CI 2-sided [104.03 to 127.34]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; [analysis description as in outcome 1, analysis 2]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 145.60, 90% CI 2-sided [131.68 to 160.99]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; [analysis description as in outcome 1, analysis 3]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 161.48, 90% CI 2-sided [145.95 to 178.66]

4. Primary Outcome: AUCinf of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: as for outcome 1
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
ng*hr/mL | 4843 (28) | 5414 (30) | 4979 (45) | 5271 (26)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; [analysis description as in outcome 1, analysis 1]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 110.85, 90% CI 2-sided [95.38 to 128.82]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; [analysis description as in outcome 1, analysis 2]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 106.55, 90% CI 2-sided [91.76 to 123.73]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; [analysis description as in outcome 1, analysis 3]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 107.74, 90% CI 2-sided [92.70 to 125.21]

5. Primary Outcome: AUClast of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: as for outcome 2
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
ng*hr/mL | 4588 (29) | 5108 (32) | 4757 (46) | 4998 (26)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; [analysis description as in outcome 1, analysis 1]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 110.19, 90% CI 2-sided [94.51 to 128.47]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; [analysis description as in outcome 1, analysis 2]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 107.17, 90% CI 2-sided [92.00 to 124.86]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; [analysis description as in outcome 1, analysis 3]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 107.83, 90% CI 2-sided [92.48 to 125.72]

6. Primary Outcome: Cmax of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles Under Fasted Conditions
Description: Maximum plasma concentration (Cmax) was measured. Cmax was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each period
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
ng/mL | 536.9 (41) | 598.2 (42) | 579.8 (45) | 640.5 (30)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water; [analysis description as in outcome 1, analysis 1]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric means = 108.72, 90% CI 2-sided [89.32 to 132.32]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce; [analysis description as in outcome 1, analysis 2]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 109.44, 90% CI 2-sided [90.05 to 133.00]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding; [analysis description as in outcome 1, analysis 3]; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of Adjusted Geometric Means = 117.30, 90% CI 2-sided [96.37 to 142.77]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Event
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product, without regard to relatedness. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Treatment-related TEAEs were any untoward medical occurrence attributed to study intervention. Relatedness to study intervention was determined by the investigator.
Time Frame: Baseline up to Follow-up (35 days after last dose administration), an average of 10 weeks.
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants
  All-causality TEAEs | 6 | 2 | 1 | 4
  Treatment-related TEAEs | 3 | 2 | 1 | 1

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants analyzed in the laboratory abnormalities were with at least one observation of the given laboratory test while on study treatment or during lag time. Number of participants with laboratory abnormalities were number of participants with a laboratory abnormality meeting specified criteria while on study treatment or during lag time. Hematology, chemistry, urinalysis and other (SARS-CoV-2 RT-PCR, Urine drug screening, Pregnancy test (β hCG), eGFR [CKD-EPI], aPTT, PT-INR, Fibrinogen, At Screening only: FSH, HBsAg, HBsAb, HBcAb, HCVAb, HIV) were assessed.
Time Frame: Screening, Period 1 Day -1, Period 4 Day 4 and early termination/discontinuation.
Population: All participants who took at least 1 dose of study intervention were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 3 | 2 | 4 | 3
Participants
  Urinalysis: pH (>8) | 0 | 1 | 0 | 0
  Urinalysis: Urine hemoglobin (≥1) | 1 | 0 | 0 | 0
  Urinalysis: Nitrite (≥1) | 0 | 1 | 0 | 0
  Urinalysis: Leukocyte Esterase (≥1) | 1 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Values
Description: Participants with clinically significant vital sign values were with at least one observation of vital signs, which met pre-specified criteria while on study treatment or during lag time.
Time Frame: Screening, Day 1 of each period and early termination/discontinuation.
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Values
Description: Participants with clinically significant physical examination values were with at least one observation of physical examination, which met pre-specified criteria while on study treatment or during lag time.
Time Frame: Screening and Period 1 Day -1.
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram Values
Description: Participants with clinically significant electrocardiogram (ECG) values were with at least one observation of ECG, which met pre-specified criteria while on study treatment or during lag time.
Time Frame: Screening, Period 1 Day 1 and Period 4 Day 4.
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Taste Assessment of Mouth Feel After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: Participants reviewed the taste questionnaire and instructions prior to the first taste assessment to treatments (B, C, D) on Period 1 Day 1. Each participant completed the Taste Assessment Survey immediately following dosing (within 1 min) and at 5, 10, and 20 minutes post oral administration of PF-07321332/ritonavir oral powder. For the taste assessment in the study, the data used in the analysis were transcribed and rescaled to a score from 0 to 100 from the raw measurements on the Taste Assessment Questionnaire. The score of 0 was considered Favorable and the score of 100 was considered Not Favorable. Higher score means more unfavorable.
Time Frame: 1, 5, 10, 20 min after tasting each study intervention on Day 1 of each period.
Population: All participants who had tasted study interventions (in different vehicles) and made scores on the taste questionnaires were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 12 | 11
Units on a scale
  1 min | 61.3 (31.25) | 53.5 (28.42) | 49.5 (31.30)
  5 min | 63.2 (36.52) | 55.2 (32.56) | 57.5 (34.18)
  10 min | 61.2 (35.96) | 52.5 (38.92) | 51.6 (37.29)
  20min | 60.5 (35.06) | 52.0 (37.26) | 48.5 (35.41)

13. Secondary Outcome: Taste Assessment of Bitterness After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 12
Time Frame: 1, 5, 10, 20 min after tasting each study intervention on Day 1 of each period.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 12 | 11
Units on a scale
  1 min | 75.4 (27.37) | 69.3 (34.39) | 63.2 (33.48)
  5 min | 76.4 (29.15) | 65.0 (35.46) | 63.2 (34.91)
  10 min | 69.8 (31.47) | 67.3 (35.16) | 64.6 (37.72)
  20min | 73.4 (32.39) | 64.7 (34.15) | 61.4 (38.49)

14. Secondary Outcome: Taste Assessment of Tongue/Mouth Burn After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 12
Time Frame: 1, 5, 10, 20 min after tasting each study intervention on Day 1 of each period.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 12 | 11
Units on a scale
  1 min | 42.5 (28.18) | 38.7 (30.57) | 31.2 (28.69)
  5 min | 45.5 (34.74) | 35.3 (30.52) | 35.0 (31.38)
  10 min | 43.7 (33.07) | 32.4 (30.46) | 37.6 (36.98)
  20min | 42.6 (35.50) | 33.8 (30.76) | 36.6 (31.50)

15. Secondary Outcome: Taste Assessment of Throat Burn After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 12
Time Frame: 1, 5, 10, 20 min after tasting each study intervention on Day 1 of each period.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 12 | 11
Units on a scale
  1 min | 37.4 (29.85) | 34.6 (32.15) | 27.6 (24.17)
  5 min | 42.6 (32.04) | 29.7 (29.61) | 34.9 (31.35)
  10 min | 40.7 (31.09) | 30.7 (29.63) | 39.5 (38.53)
  20min | 40.5 (33.32) | 32.5 (29.41) | 40.3 (35.70)

16. Secondary Outcome: Taste Assessment of Overall Liking After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 12
Time Frame: 1, 5, 10, 20 min after tasting each study intervention on Day 1 of each period.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
Number analyzed (Participants) | 11 | 12 | 11
Units on a scale
  1 min | 77.9 (28.53) | 62.5 (33.89) | 61.8 (34.69)
  5 min | 78.2 (30.28) | 67.0 (34.27) | 66.5 (38.34)
  10 min | 77.9 (30.83) | 67.5 (37.16) | 64.6 (38.99)
  20min | 75.2 (32.14) | 65.0 (35.98) | 63.9 (40.19)

ADVERSE EVENTS:
Time Frame: Baseline up to Follow-up (35 days after last dose administration), an average of 10 weeks.
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 2/11 | 1/12 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir/Ritonavir 300/100 mg Commercial Tablets (N=11) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (N=11) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Applesauce (N=12) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (N=11)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT05263921/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT05263921/SAP_001.pdf